CLINICAL TRIAL: NCT01684137
Title: Monitoring of Allergic and Asthmatic Symptoms in Patients Taking Dietary Supplements Joalis Bambi Bronchi and Joalis Bambi Analerg
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: DSC Services, s.r.o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: KS-2011-05-JOALIS
Record Dates: First submitted 2012-08-21; First posted 2012-09-12 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Children
Keywords: Food supplements; Asthma bronchiale

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Joalis Bambi Bronchi & Joalis Bambi Analerg (Active Comparator): 10 days, 2 times per day 2,5/5 ml
  Interventions: Dietary Supplement: Joalis Bambi Analerg; Dietary Supplement: Joalis Bambi Bronchi
- Placebo & Placebo (Placebo Comparator): 10 days, 2 times per day 2,5/5 ml
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Joalis Bambi Analerg
  Arms: Joalis Bambi Bronchi & Joalis Bambi Analerg
Dietary Supplement: Joalis Bambi Bronchi
  Arms: Joalis Bambi Bronchi & Joalis Bambi Analerg
Dietary Supplement: Placebo — Sugar pill manufactured to mimic Joalis Bambi Analerg
  Arms: Placebo & Placebo
Dietary Supplement: Placebo — Sugar pill manufactured to mimic Joalis Bambi Bronchi
  Arms: Placebo & Placebo

SUMMARY:
Reduction of the total IgE antibody, improved vital capacity and lung volume measured by spirometry.

Improving quality of life observed in the visual analogue scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* subjects with confirmed Asthma bronchiale I-III. degrees in possible combination with other allergic symptoms treating with classic pharmacological treatment
* 9-18 years
* signed Infromed Conset

Exclusion Criteria:

* subjects who have previously used a food suplemts Joalis
* subjects with known intolerance or hypersensitivity to the components of food supplements
* subjects with alcohol abuse or drugs at the time of recruitment into the study
* subjects enrolled in another clinical trial in the last 1 month before enrollment in this study
* subjects in a situation which in the opinion of a doctor may interfere with optimal participation in the study or can pose a risk to the subjects
* pregnant girls, lactating girls and girls of childbearing age without adequate contraception

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Reduction of the total IgE (IU/ml) antibody. | 1 year
Improving of vital capacity measured by spirometry (litre). | 1 year
Improving of lung volume measured by spirometry (litre). | 1 year

SECONDARY OUTCOMES:
Improving of quality of life observed in the visual analogue scale (VAS). | 1 year

OTHER OUTCOMES:
Asthma bronchiale, age 9-18 year | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Karel Chroust, RNDr., Ing., PhD., Study Director — DSC Services, s.r.o.
Locations (1):
- Alergologická ambulance, Zlín, Czechia